CLINICAL TRIAL: NCT02920437
Title: A Pilot Randomized Controlled Trial to Reduce Salt Intake Among Hypertensive Young Adults in Hong Kong
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study cannot recruit the expected number of participants. Only 19 participants were recruited and no more new participant was recruited after that.
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Pui-Hing Chau, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 16-280
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Hypertension
Keywords: dietary salt; 24 hour urinary sodium excretion; blood pressure; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Four-week weekly intervention to reduce salt intake.
  Interventions: Behavioral: Four-week weekly intervention to reduce salt intake
- Control group (Other): Usual government pamphlets.
  Interventions: Other: Usual government pamphlets

INTERVENTIONS:
Behavioral: Four-week weekly intervention to reduce salt intake — The intervention group will receive a four-week weekly intervention, about 15 minutes each. Two sessions will be face-to-face and two sessions will be on the phone. The participants will be informed of their 24-hour urinary sodium excretion at each measurement time once available.
  Arms: Intervention group
Other: Usual government pamphlets — The control group will receive usual government pamphlets when they know their 24-hour urinary sodium excretion at baseline. However, they will not be informed of their follow-up urinary sodium excretion results immediately.
  Arms: Control group

SUMMARY:
A pilot randomized controlled trial will be conducted to investigate the feasibility and effectiveness of a salt intake reduction intervention to young hypertension patients in Hong Kong who had high salt intake.

DETAILED DESCRIPTION:
Convenience sample will be recruited from the community in Hong Kong through different channels of promotion.

ELIGIBILITY:
Inclusion Criteria:

* i) adults aged 18 to 44
* ii) diagnosed hypertension or borderline hypertension
* iii) complete collection of 24-hour urine at baseline
* iv) 24-hour urinary sodium excretion above 2000mg at baseline
* v) can communicate in Cantonese

Exclusion Criteria:

* i) renal illnesses;
* ii) taking diuretics;
* iii) taking RAS blockers;
* iv) attending or planning to attend new hypertension education programme or salt intake reduction programme during the study period.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
24-hour urinary sodium excretion | 10-Week
  Difference between the intervention and control group in the change in 24-hour urinary sodium excretion from baseline to the end of follow-up

SECONDARY OUTCOMES:
Health literacy on low salt intake | 10-Week
  Difference between the intervention and control group in the change in health literacy on low salt intake measured with the validated Chinese Health Literacy Scale for Low Salt Consumption (CHLSalt-HK)

CONTACTS AND LOCATIONS:
Overall Officials: Chau Pui Hing, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No